CLINICAL TRIAL: NCT02882282
Title: Personalized, Randomized, Phase 2 Study of Pembrolizumab (MK-3475) for High Risk Oral Intra-Epithelial Neoplasias
Brief Title: Pembrolizumab in Treating Patients With High Risk Oral Intraepithelial Neoplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0193; NCI-2017-00479 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0193 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-08-24; First posted 2016-08-29 (Estimated); Results first posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-08

CONDITIONS: Oral Cavity Carcinoma; Oral Intraepithelial Neoplasia
MeSH Terms: conditions — Mouth Neoplasms | interventions — Watchful Waiting; Observation; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (observation) (Active Comparator): Patients undergo observation.
  Interventions: Other: Patient Observation
- Arm B (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
  Arms: Arm B (pembrolizumab)
Other: Patient Observation — Undergo observation
  Other Names: Active Surveillance; deferred therapy; expectant management; Observation; watchful waiting
  Arms: Arm A (observation)
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
  Arms: Arm B (pembrolizumab)

SUMMARY:
This randomized phase II trial studies how well pembrolizumab works in treating patients with high risk oral intraepithelial neoplasia. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine oral cancer-free survival of patients with high risk oral intra-epithelial neoplasias (IEN) treated with pembrolizumab versus observation.

SECONDARY OBJECTIVES:

I. To determine the safety and tolerability of pembrolizumab for patients with oral IEN.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients undergo observation.

ARM B: Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 6, 9, 12, 18, 24, 30, and 36 months and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histological evidence of oral intra-epithelial neoplasia within 12 months prior to enrollment; subjects with a history or clinical diagnosis suggestive of oral intra-epithelial neoplasia, or patients with a history of invasive oral cancer are eligible, but must have a confirmed histological diagnosis of oral intra-epithelial neoplasia before randomization; histological evidence of oral intraepithelial neoplasia on an invasive oral cancer resection specimen is acceptable; a visible, measurable, clinical lesion (such as leukoplakia and/or erythroplakia) is not required; only individuals with high risk profiles will be considered eligible for randomization; high risk profiles are defined as patients without a prior oral cancer and have loss of heterozygosity (LOH) at 3p14 and/or 9p21 plus at least at one additional chromosomal site (4q,8p,11p,13q, or 17p) or patients with a prior oral cancer history and have LOH at 3p14 and/or 9p21; all high risk patients must also meet the additional eligibility criteria
* Be willing and able to provide written informed consent
* Be greater than or equal to 18 years of age on day of signing informed consent for the trial
* Be willing to provide tissue from a newly obtained oral biopsy
* Have a performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 75,000/mcL
* Serum total bilirubin =< 1.5 X upper limit of normal (ULN) or direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN
* Female subject of childbearing potential should have a negative urine or serum pregnancy test < 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of study therapy through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses > 1 year
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of the study therapy

Exclusion Criteria:

* Is currently participating and receiving study therapy with potential anti-neoplastic activity, or has participated in a study of an investigational agent and received study therapy with potential anti-neoplastic activity within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has a known history of active TB (Bacillus tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 2 at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 2 or at baseline) from adverse events due to a previously administered agent; Note: If the subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment other than adjuvant hormonal therapy; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin or in situ cervical cancer
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has a known history of, or any evidence of active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant, or breastfeeding, or expecting to conceive or father children within the projected duration of treatment with pembrolizumab, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Has a history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days of planned start of study therapy; Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renata Ferrarotto, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Control): Observation
- Arm B (Pembrolizumab).: Pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 4 courses until disease progression or unacceptable toxicity
Period: Overall Study
Arm/Group | Arm A (Control) | Arm B (Pembrolizumab).
Started | 7 | 8
Completed | 7 | 7
Not Completed | 0 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Control) | Arm B (Pembrolizumab) | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 3 | 4 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 | 9
  Male | 5 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 7 | 14
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Oral Cancer-free Survival
Description: To determine oral cancer-free survival and overall survival of patients with high risk oral IEN treated with Pembrolizumab versus observation
Time Frame: 51.2 months
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Arm B (Pembrolizumab ): Pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 4 courses until disease progression or unacceptable toxicity
Arm/Group | Arm A (Control) | Arm B (Pembrolizumab )
Number analyzed (Participants) | 7 | 8
Months | NA [NA to NA] — Not reached | 6.7 [3.6 to 40.2]

2. Secondary Outcome: Overall Survival
Description: To determine overall survival of patients with high risk oral IEN treated with pembrolizumab versus observation. The distribtuion of overall survival was estimated using Kaplan-Meier method.
Time Frame: Overall survival was defined as from the randomization to death of all causes, whichever occurred first or last follow up.
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Control) | Arm B (Pembrolizumab).
Number analyzed (Participants) | 7 | 8
months | NA [NA to NA] — Not reached | NA [NA to NA] — Not reached

ADVERSE EVENTS:
Time Frame: Approximately 4 years, 4 months
Groups:
- Arm A: Observation (Control)
- Arm B: Pembrolizumab 4 doses (experimental)
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 1/7 | 7/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 6/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=7) | Arm B (N=8)
Constipation (Gastrointestinal disorders) | 0 | 4
Fatigue (General disorders) | 0 | 3
Mucositis Oral (Gastrointestinal disorders) | 0 | 2
Hypothyroidism (General disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Non-Cardiac chest pain (Gastrointestinal disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Chest Pain - Cardiac (Cardiac disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Ear Pain (General disorders) | 0 | 1
Flu Like Symptoms (General disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hot flashes (Vascular disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Joint Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Oral secretion (Gastrointestinal disorders) | 0 | 1
Peg Placement (Gastrointestinal disorders) | 0 | 1
Rash pustular (Infections and infestations) | 0 | 1
sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
vomiting (Gastrointestinal disorders) | 0 | 1
White blood cell decreased (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-09): https://cdn.clinicaltrials.gov/large-docs/82/NCT02882282/Prot_SAP_001.pdf